CLINICAL TRIAL: NCT03652779
Title: An Open-label, Phase 1, Sequential Cohort, Single-Dose Escalation Study to Assess the Safety and Tolerability of Tecarfarin (ATI-5923) in Healthy Chinese Volunteers
Brief Title: A Study to Evaluate the Safety and Tolerability of Tecarfarin in Healthy Chinese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: LP-HK-001
Record Dates: First submitted 2018-08-28; First posted 2018-08-29 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-09

CONDITIONS: Pharmacokinetic and Pharmacodynamic Profile of Tecarfarin
MeSH Terms: interventions — tecarfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tecarfarin 10mg (Experimental)
  Interventions: Drug: Tecarfarin 10mg
- Tecarfarin 20mg (Experimental)
  Interventions: Drug: Tecarfarin 20mg
- Tecarfarin 30mg (Experimental)
  Interventions: Drug: Tecarfarin 30mg
- Tecarfarin 40mg (Experimental)
  Interventions: Drug: Tecarfarin 40mg

INTERVENTIONS:
Drug: Tecarfarin 10mg — Tecarfarin 10mg tablets
  Arms: Tecarfarin 10mg
Drug: Tecarfarin 20mg — two tecarfarin 10mg tablets
  Arms: Tecarfarin 20mg
Drug: Tecarfarin 30mg — three tecarfarin 10mg tablets
  Arms: Tecarfarin 30mg
Drug: Tecarfarin 40mg — four tecarfarin 10mg tablets
  Arms: Tecarfarin 40mg

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of a single dose of tecarfarin in healthy Chinese Volunteers. the Pharmacokinetic and pharmacodynamic profile of tecarfarin will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must voluntarily sign and date an informed consent form, approved by the Institutional Review Board (IRB), prior to the initiation of any study-specific procedure.
2. Healthy Chinese* volunteers aged between 18 and 55 years inclusive, at the time of Screening

   *Definition of "Chinese": Subject is a Han Chinese who born in China (including Hong Kong) with Han Chinese parents and grandparents who born in China (including Hong Kong).
3. Body Mass Index (BMI) ≥19 and ≤ 24 kg/m2
4. Subject has been a non-smoker or has not used tobacco or nicotine-containing products for at least 3 months before Screening and prior to Day 1.
5. Subjects are in general good health with no history of significant diseases and no clinically significant abnormal findings based upon the results of physical examination, 12-lead ECG, laboratory safety tests and vital signs at screening and prior to dosing.

   • Vital signs (measured in a sitting position for at least 5 minutes) include tympanic temperature [T], pulse rate [PR], respiratory rate [RR], and blood pressure [BP]).
6. Female subjects must be non-pregnant, non-lactating or either postmenopausal for at least 2 years or surgically sterile (e.g., hysterectomy, bilateral oophorectomy, bilateral tubal occlusion or ligation) for at least 6 months. For female subjects of child bearing potential, they need to consentient to use appropriate contraceptive methods (abstinence, intrauterine device, diaphragm with spermicide, use by partner of a condom with spermicide) at least 28 days prior to and after dosing. Use of oral contraceptive and implantation of contraceptive methods by female subjects are not acceptable.
7. Male subjects who have female partners of reproductive potential must either:

   * Abstinence from sexual intercourse during Day -1 to Day 28, or
   * Use an approved method of contraception (which may include use of a condom with spermicide or use by partner of oral, implantable or injectable contraceptives, intrauterine device, diaphragm with spermicide) during Day -1 to Day 28.
   * Refrain from sperm donation during Day -1 to Day 28.
8. Able and willing to follow instructions and to comply with protocol requirements.

Exclusion Criteria:

1. Positive test results for HIV, syphilis antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody (HCV Ab) at Screening.
2. Positive tests for alcohol breathalyzer or urine drugs of abuse at Screening or Day -1 or a history of drug abuse/dependence.
3. Use of tobacco or nicotine products 3 months before screening and prior to Day 1.
4. Heavy caffeine drinker (> 5 cups or glasses of caffeinated beverages [e.g., coffee tea, cola, energy drinks] per day) within 3 months prior to screening.
5. Heavy alcohol drinker (more than 30 gram alcohol per day within 3 months prior to screening (30 gram alcohol is approximately equivalent to: i.e. 100ml of aperitif, 300ml of wine or 500ml of beer)).
6. Any clinically significant above normal range of prothrombin time, activated partial thromboplastin time, or international normalized ratio or below normal range of Protein C or Protein S laboratory result at Screening.
7. Documented history of bleeding diathesis, coagulopathy, or inherited disorders of coagulation.
8. Evidence of active bleeding, including but not limited to bleeding ulcer, bleeding gums, urinalysis positive for more than trace blood at Screening and presence of occult blood in the stool at Screening.
9. Subjects with a QTcB interval (QT interval corrected for heart rate according to Bazett's formula) > 450 msec at Screening, confirmed by a repeat assessment.
10. Conditions predisposing to QT prolongation including pathological Q-wave (defined as Q-wave >40 msec or depth > 0.4-0.5 mV).
11. History or presence of cardiac abnormalities or congenital long QT syndrome based on the final investigators' judgment.
12. History or presence of malignancy within the past 2 years, with the exception of adequately treated localized skin cancer (basal cell or squamous cell carcinoma) or carcinoma in-situ of the cervix.
13. Participation in a previous clinical trial within 3 months prior to Screening.
14. Clinically significant surgical procedure within 3 months prior to Screening.
15. Clinically significant blood loss or blood donation > 550 ml within 3 months prior to Day 1.
16. Any laboratory results from complete blood picture suspicious of ongoing blood loss.
17. Taking any prescription medication 14 days prior to Day -1.
18. Routine or as needed consumption of medications, herbal, vitamins or hormone supplements 14 days prior to Day -1 or subject is unable to withhold these medications due to underlying clinical conditions, or unwilling to refrain from taking these medications, during the study period (Day -1 to Day 15).
19. Known allergy or hypersensitivity to warfarin or the investigational product.
20. Any other conditions or clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during Screening that, in the opinion of the Principal Investigator would make the subject unsuitable for the study or put them at additional risks.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2019-10-28 (Actual)

PRIMARY OUTCOMES:
Adverse Events Frequency | 15 Days
Adverse Events Severity | 15 Days

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve | 336 Hours
Peak Plasma Concentration | 336 Hours
Time which Peak Plasma Concentration is Reached | 336 Hours
Elimination Rate Constant | 336 Hours
Elimination Half Life | 336 Hours
Clearance | 336 Hours
Volume of Distribution | 336 Hours
International Normalized Ratios | 0 hour, 1 hour, 4 hours, 8 hours,12 hours, day 2, day 3, day 4, day 8, day 15
Prothrombin Time | 0 hour, 1 hour, 4 hours, 8 hours,12 hours, day 2, day 3, day 4, day 8, day 15
Activated Partial Thromboplastin Time | 0 hour, 1 hour, 4 hours, 8 hours,12 hours, day 2, day 3, day 4, day 8, day 15
Coagulation Factor II | 8 Days
  0 hour, 1 hour, 4 hours, 8 hours,12 hours, day 2, day 3, day 4, day 8, day 15
Coagulation Factor VII | 8 Days
  0 hour, 1 hour, 4 hours, 8 hours,12 hours, day 2, day 3, day 4, day 8, day 15
Coagulation Factor X | 8 Days
  0 hour, 1 hour, 4 hours, 8 hours,12 hours, day 2, day 3, day 4, day 8, day 15

CONTACTS AND LOCATIONS:
Overall Officials: Jo Jo SH Hai, MBBS, Principal Investigator — Queen Mary Hospital, Hong Kong
Locations (1):
- HKU Phase 1 Clinical Trial Centre, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No